CLINICAL TRIAL: NCT03438474
Title: Pelvic and Para-aortic Lymphadenectomy in Patients With Stage I or II Endometrial Cancer With High Risk of Recurrence
Brief Title: Endometrial Cancer Lymphadenectomy Trial
Acronym: ECLAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: German Cancer Aid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OP.6 KKS 228
Record Dates: First submitted 2018-01-31; First posted 2018-02-19 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Cancer of Endometrium Stage I; Cancer of Endometrium Stage II
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A standard surgical procedure (Active Comparator): Standard surgical procedure for endometrial cancer:
  total hysterectomy, bilateral salpingo-oophorectomy, omentectomy (type 2 cancers)
  Interventions: Procedure: Standard surgical procedure for endometrial cancer
- Arm B systematic lymphadenectomy (LNE) (Experimental): In addition to standard procedures as defined for Arm A:
  systematic pelvic and para-aortic lymphadenectomy (LNE) up to the renal vessels
  Interventions: Procedure: Standard surgical procedure for endometrial cancer; Procedure: systematic lymphadenectomy (LNE)

INTERVENTIONS:
Procedure: Standard surgical procedure for endometrial cancer — total hysterectomy, bilateral salpingo-oophorectomy, omentectomy (type 2 cancers)
Procedure: systematic lymphadenectomy (LNE) — systematic pelvic and para-aortic lymphadenectomy (LNE) up to the renal vessels
  Arms: Arm B systematic lymphadenectomy (LNE)

SUMMARY:
The primary aim of this trial is to ascertain whether or not systematic pelvic and para-aortic lymphadenectomy (LNE) does have a significant impact on overall survival (OS) in patients with endometrial cancer (EC) FIGO Stages I or II and high risk of recurrence. Secondary aims will be to evaluate the effect of LNE on disease free survival (DFS) and quality of life, as well as the complications and side effects of LNE and the number of resected lymphnodes. 640 patients with histologically confirmed EC with high risk of recurrence (stage pT1b - pT2, all histological subtypes; pT1a, G3 endometrioid or serous or clear cell EC or carcinosarcomas) will be randomized. In Arm A, a total hysterectomy and bilateral salpingo-oophorectomy and in case of serous or clear cell EC additionally an omentectomy will be performed. In arm B in addition a systematic pelvic and para-aortic LNE up to the level of the left renal vein will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed EC of clinical stages T1b and T2 (all histological types) and stage T1a G3 type 1 (endometrioid, endometriod with squamous differentiation, mucinous) or type 2 tumors (any percentage of serous or clear cell component) or carcinosarcoma
2. a) no previous surgery concerning EC (primary surgery) or b) surgery after hysterectomy (e.g. for presumed low risk endometrial cancer) is allowed within 8 weeks after hysterectomy if no LNE was performed (secondary surgery)
3. absence of bulky lymph nodes
4. performance status ECOG 0-1
5. age 18 - 75 years
6. written informed consent
7. adequate compliance

Exclusion Criteria:

1. stage pT1a, G1 or G2 tumors of type 1 histology
2. sarcomas (except for carcinosarcoma = malignant mixed Müllerian tumor)
3. EC of FIGO stages III or IV (except for microscopical lymph node metastases)
4. evidence of extrauterine disease by visual inspection
5. recurrent EC
6. preceding chemo-, radio, or endocrine therapy for EC
7. any concomitant disease not allowing surgery including lymphadenectomy and/or chemotherapy
8. any medical history indicating excessive peri-operative risk
9. any current medication containing considerable surgical risk (e.g. bleeding: due to oral anticoagulating agents)
10. any known disorder or circumstances making participation in trial and follow-up questionable. Insufficient compliance is expected.
11. patients with second malignancies if disease or treatment might have an impact on the patient's prognosis
12. known HIV-infection or AIDS
13. simultaneous participation in other clinical trials if not permitted by the steering committee (translational or QoL studies not interfering with the objectives of ECLAT are allowed)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2028-02-15 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 60 months
  Impact of systematic pelvic and para-aortic lymphadenectomy (LNE) on overall survival in EC patients with high risk of recurrence

SECONDARY OUTCOMES:
Disease free survival (DFS) | 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months, 27 months, 30 months, 33 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Impact of systematic pelvic and para-aortic lymphadenectomy (LNE) on Disease free survival
Disease specific survival (DSS) | 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months, 27 months, 30 months, 33 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Impact of systematic pelvic and para-aortic lymphadenectomy (LNE) on Disease specific survival
Assessment of serious complications | during surgery, at hospital discharge, day 60, 6 months, 9 months, 12 months
  Assessment of perioperative complications and site effects of LNE
EORTC QLQ-C30 | Baseline, at hospital discharge, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months, 27 months, 30 months, 33 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Health related Quality of life (QoL)
EORTC QLQ-EN24 | Baseline, at hospital discharge, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months, 27 months, 30 months, 33 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Health related Quality of life (QoL)
Number of resected lymph nodes | during surgery
  resected pelvic and para-aortic lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Harter, Professor MD, Principal Investigator — Kliniken Essen Mitte, Gynäkologie und gynäkologische Onkologie
Locations (61):
- Germany (58):
  - Ostalb-Klinikum Aalen, Frauenklinik, Aalen
  - Klinikum St. Marien Amberg, Frauenklinik, Amberg
  - Klinikum Ansbach, Klinikum Ansbach, Ansbach
  - Universitätsklinikum Augsburg, Frauenklinik, Augsburg
  - Hochtaunus-Kliniken gGmbH, Frauenklinik, Bad Homburg
  - Sozialstiftung Bamberg, Klinikum am Bruderwald, Klinik für Frauenheilkunde, Bamberg
  - SANA Klinikum Lichtenberg, Oskar-Ziehten-Krankenhaus, Frauenklinik, Berlin
  - Vivantes Auguste-Viktoria-Klinikum, Klinik für Gynäkologie und Geburtsmedizin, Berlin
  - Charité Campus Virchow-Klinikum, Klinik für Frauenheilkunde und Geburtshilfe, Berlin
  - Vivantes Humboldt-Klinikum, Klinik für Gynäkologie und Geburtsmedizin, Berlin
  - Martin-Luther-Krankenhaus, Klinik für Gynäkologie und Geburtshilfe, Berlin
  - Universitätsklinikum Bonn, Zentrum für Geburtshilfe u. Frauenheilkunde, Bonn
  - Sana Kliniken Leipziger Land GmbH, Klinik für Gynäkologie und Geburtshilfe, Borna
  - Kliniken Böblingen, Frauenklinik, Böblingen
  - Städtisches Klinikum Braunschweig gGmbH, Frauenklinik, Braunschweig
  - Klinikum Bremen Mitte gGmbH, Frauenklinik, Bremen
  - Evangelisches Krankenhaus Kalk gGmbH, Gynäkologie und Geburtshilfe, Cologne
  - Donau-Ries Klinik Donauwörth, Klinik für Frauenheilkunde und Geburtshilfe, Donauwörth
  - Universitätsklinikum Carl Gustav Carus, Klinik u. Poliklinik f. Frauenheilkunde u. Geburtshilfe, Dresden
  - Kaiserswerther-Diakonie, Florence-Nightingale-Krankenhaus, Gynäkologie u. Geburtshilfe, Düsseldorf
  - Kliniken Essen Mitte, Evang. Huyssens Stiftung/Knappschaft GmbH, Gynäkologische Onkologie, Essen
  - Klinikum der Johann Wolfgang Goethe Universität, Klinik für Gynäkologie und Geburtshilfe, Frankfurt am Main
  - Universitätsklinikum Freiburg, Universitätsfrauenklinik, Freiburg im Breisgau
  - Klinikum Fulda gAG, Frauenklinik, Fulda
  - Klinikum Fürth, Frauenklinik Nathanstift, Fürth
  - Universitätsklinikum Gießen und Marburg GmbH, Frauenklinik, Giessen
  - Klinikum Göttingen, Georg-August-Universität, Universitätsfrauenklinik, Göttingen
  - Klinikum der Ernst-Moritz-Arndt-Universität, Klinik u. Poliklinik f. Gynäkologie u. Geburtshilfe, Greifswald
  - Klinikum Gütersloh, Frauenklinik, Gütersloh
  - Universitätsklinikum Halle/S., Universitätsklinik und Poliklinik für Gynäkologie, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Klinik und Poliklinik für Gynäkologie, Hamburg
  - Agaplesion Diakonieklinikum Hamburg, Frauenklinik, Hamburg
  - Albertinen Krankenhaus/Albertinen-Haus gemeinnützige GmbH, Station B2 Gynäkologie, Hamburg
  - Medizinische Hochschule Hannover, Frauenklinik, Hanover
  - Universitätsklinikum Jena, Klinik für Frauenheilkunde und Geburtshilfe, Jena
  - Städtisches Klinikum Karlsruhe, Frauenklinik, Karlsruhe
  - ViDia Christliche Kliniken Karlsruhe, Frauenklinik, Karlsruhe
  - Klinikum Mannheim GmbH, Universitäts-Frauenklinik, Mannheim
  - Evangelisches Krankenhaus Bethesda, Klinik für Frauenheilkunde und Geburtshilfe, Mönchengladbach
  - Klinikum Dritter Orden, Klinik für Gynäkologie und Geburtshilfe, München
  - Klinikum der Universität München (LMU), Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, München
  - Klinikum rechts der Isar der Technischen Universität, Frauen- und Poliklinik, München
  - Klinikum Offenbach GmbH, Frauenklinik, Offenbach
  - Ortenau Klinikum St. Josefsklinik, Gynäkologie, Offenburg
  - Klinikum Passau, Frauenklinik, Passau
  - Oberschwabenklinik Krankenhaus St. Elisabeth, Frauenklinik, Ravensburg
  - Caritas-Krankenhaus St. Josef, Klinik für Frauenheilkunde u. Geburtshilfe, Regensburg
  - Leopoldina Krankenhaus Schweinfurt GmbH, Frauenheilkunde und Geburtshilfe, Schweinfurt
  - Städt. Klinikum Solingen gGmbH, Frauenheilkunde u. Geburtshilfe, Solingen
  - Klinikum Starnberg, Klinik für Frauenheilkunde und Geburtshilfe, Starnberg
  - Klinikum St. Elisabeth Straubing GmbH, Klinik für Frauenheilkunde und Geburtshilfe, Straubing
  - Kreiskliniken Traunstein-Trostberg GmbH, Frauenklinik, Traunstein
  - Universitätsklinikum Tübingen, Universitätsfrauenklinik, Tübingen
  - Universitätsklinikum Ulm, Universitätsfrauenklinik, Ulm
  - Christliches Klinikum Unna Mitte, Klinik für Gynäkologie und Geburtshilfe, Unna
  - Schwarzwald-Baar Klinikum, Frauenklinik, Villingen-Schwenningen
  - St. Josefs-Hospital, Frauenklinik, Wiesbaden
  - Klinikum der Stadt Wolfsburg, Frauenklinik, Wolfsburg
- Japan (2):
  - Okayama University Hospital, Okayama
  - Saitama Medical University International Medical Center, Saitama
- Seoul National University Hospital, Department of Obstetrics & Gynecology, Seoul, South Korea

REFERENCES:
- [Derived] Emons G, Kim JW, Weide K, de Gregorio N, Wimberger P, Trillsch F, Gabriel B, Denschlag D, Kommoss S, Aydogdu M, Papathemelis T, Gropp-Meier M, Muallem MZ, Kuhn C, Muller A, Frank M, Weigel M, Bronger H, Lampe B, Rau J, Schade-Brittinger C, Harter P. Endometrial Cancer Lymphadenectomy Trial (ECLAT) (pelvic and para-aortic lymphadenectomy in patients with stage I or II endometrial cancer with high risk of recurrence; AGO-OP.6). Int J Gynecol Cancer. 2021 Jul;31(7):1075-1079. doi: 10.1136/ijgc-2021-002703. PMID 34226291